CLINICAL TRIAL: NCT06594003
Title: Comparative Study Between Eight Versus Three Genicular Nerves Radiofrequency Ablation for Knee Denervation in Advanced Knee Osteoarthritis Using Ultrasound
Brief Title: Motor Sparing Techniques, Genicular Nerve Radiofrequency Ablation Has Emerged As a Viable Alternative to Conservative Therapy and Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Ibrahim Mubarak, teaching assistant, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: genicular nerves ablation
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis (OA)
Keywords: knee; osteoarthritis; radiofrequency; genicular nerves
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- three genicular nerves raiofrequency ablation (Active Comparator)
  Interventions: Procedure: Radiofrequency
- eight genicular nerves radiofrequency ablation (Active Comparator)
  Interventions: Procedure: Radiofrequency

INTERVENTIONS:
Procedure: Radiofrequency — There has recently been considerable interest in the role of radiofrequency ablation (RFA) of the genicular nerves for KOA. In the majority of previous studies, ablation was done via a radiofrequency technique using either fluoroscopy or ultrasound for only three genicular nerves, whereas the knee joint is also supplied by a few other nerves . Interestingly, neurolytic agents can also be used to ablate the nerves, and are readily available, less costly, and need less logistic support

SUMMARY:
There has recently been considerable interest in the role of radiofrequency ablation (RFA) of the genicular nerves for KOA. In the majority of previous studies, ablation was done via a radiofrequency technique using either fluoroscopy or ultrasound for only three genicular nerves, whereas the knee joint is also supplied by a few other nerves (11, 12). Interestingly, neurolytic agents can also be used to ablate the nerves, and are readily available, less costly, and need less logistic support

DETAILED DESCRIPTION:
Knee pain is a common issue in adults, with a steadily increasing prevalence (1). There are many causes of knee pain, such as meniscal and tendon injuries, posttraumatic syndrome, and postsurgical pain; osteoarthritis is the leading cause (2).

Knee osteoarthrosis (KOA) is a very common joint disease, with a prevalence ranging from 4.2% to 15.5% and gradually increasing with age (3). It is associated with diverse causes including age, obesity, metabolic bone diseases, and acute or chronic joint injuries. Pain and disabilities are the major consequences of KOA, with 25% of patients suffering from severe arthralgia. KOA is believed to be a result of the failure of chondrocytes to maintain homeostasis between the synthesis and degradation of the extracellular matrix and from subchondral bone developing osteoarthrosis (4, 5).

Although traditional treatment modalities, including analgesics, physical therapy, and intra-articular steroid (IAS) injections, have long been employed to manage symptoms, the growing need for more effective and minimally invasive interventions has prompted the exploration of novel approaches (6).

Among these newer treatments, motor sparing techniques, genicular nerve radiofrequency ablation has emerged as a viable alternative to conservative therapy and total knee arthroplasty (7).

Genicular nerve ablation is a known procedure to help these cases as they transfer the pain signal of the knee. It is usually reserved for patients with symptomatic knee osteoarthritis who have had failure of conservative treatment and have had failure of or are poor candidates for surgery (8).

However, there is a high failure rate among the patients undergoing the procedure as regarding the efficacy or the duration of pain relief and various methods have been used to increase the rate of success and the duration of the pain relief such as using alcohol in the ablation, cooled radiofrequency or increase the lesions on the nerves (9, 10).

There has recently been considerable interest in the role of radiofrequency ablation (RFA) of the genicular nerves for KOA. In the majority of previous studies, ablation was done via a radiofrequency technique using either fluoroscopy or ultrasound for only three genicular nerves, whereas the knee joint is also supplied by a few other nerves (11, 12). Interestingly, neurolytic agents can also be used to ablate the nerves, and are readily available, less costly, and need less logistic support (13).

ELIGIBILITY:
Inclusion Criteria:

* Age from 50-70 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Patients with 3rd and 4th degree of KOA pain who undergo knee articular branch denervation via RF ablation.

Exclusion Criteria:

* Deformities in knee.
* Charcot joint (stiff Joint)
* Acute knee injury
* Previous ipsilateral total knee arthroplasty or radiofrequency denervation.
* Instability of knee Joint.
* Knee effusion & Baker's cyst . . Inability to assume a recumbent or semirecumbent position.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
vas score | 4 weeks
  will be assessed at 0, 1, and 4 weeks. on the Visual Analogue Scale (VAS) (0 = no pain, 10 = unbearable pain).

SECONDARY OUTCOMES:
Total WOMAC score. | 4 weeks
  will be assessed at 0, 1, and 4 weeks
seven-point Likert scale | 4 weeks
  seven-point Likert scale (one = worst ever, two = much worse, three = worse, four = not improved but not worse, five = improved, six = much improved, and seven = best ever).
analgesic request | 4 weeks
adverse effects | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwon HJ, Kim CS, Kim DH, Shin JW, Choi D, Choi SS. Effectiveness of the Cooled Radiofrequency Ablation of Genicular Nerves in Patients with Chronic Knee Pain Due to Osteoarthritis: A Double-Blind, Randomized, Controlled Study. Medicina (Kaunas). 2024 May 24;60(6):857. doi: 10.3390/medicina60060857. PMID 38929474
- [Background] Dass RM, Kim E, Kim HK, Lee JY, Lee HJ, Rhee SJ. Alcohol neurolysis of genicular nerve for chronic knee pain. Korean J Pain. 2019 Jul 1;32(3):223-227. doi: 10.3344/kjp.2019.32.3.223. PMID 31257831
- [Background] Wehling P, Evans C, Wehling J, Maixner W. Effectiveness of intra-articular therapies in osteoarthritis: a literature review. Ther Adv Musculoskelet Dis. 2017 Aug;9(8):183-196. doi: 10.1177/1759720X17712695. Epub 2017 Jun 20. PMID 28835778
- [Background] Kidd VD, Strum SR, Strum DS, Shah J. Genicular Nerve Radiofrequency Ablation for Painful Knee Arthritis: The Why and the How. JBJS Essent Surg Tech. 2019 Mar 13;9(1):e10. doi: 10.2106/JBJS.ST.18.00016. eCollection 2019 Mar 26. PMID 31333900
- [Background] Karm MH, Kwon HJ, Kim CS, Kim DH, Shin JW, Choi SS. Cooled radiofrequency ablation of genicular nerves for knee osteoarthritis. Korean J Pain. 2024 Jan 1;37(1):13-25. doi: 10.3344/kjp.23344. PMID 38155108
- [Background] Geng R, Li J, Yu C, Zhang C, Chen F, Chen J, Ni H, Wang J, Kang K, Wei Z, Xu Y, Jin T. Knee osteoarthritis: Current status and research progress in treatment (Review). Exp Ther Med. 2023 Aug 25;26(4):481. doi: 10.3892/etm.2023.12180. eCollection 2023 Oct. PMID 37745043
- [Background] Primorac D, Molnar V, Matisic V, Hudetz D, Jelec Z, Rod E, Cukelj F, Vidovic D, Vrdoljak T, Dobricic B, Anticevic D, Smolic M, Miskulin M, Cacic D, Boric I. Comprehensive Review of Knee Osteoarthritis Pharmacological Treatment and the Latest Professional Societies' Guidelines. Pharmaceuticals (Basel). 2021 Mar 2;14(3):205. doi: 10.3390/ph14030205. PMID 33801304
- [Background] Primorac D, Molnar V, Rod E, Jelec Z, Cukelj F, Matisic V, Vrdoljak T, Hudetz D, Hajsok H, Boric I. Knee Osteoarthritis: A Review of Pathogenesis and State-Of-The-Art Non-Operative Therapeutic Considerations. Genes (Basel). 2020 Jul 26;11(8):854. doi: 10.3390/genes11080854. PMID 32722615
- [Background] Ng TK, Lam KHS, Allam AE. Motor-Sparing Neural Ablation with Modified Techniques for Knee Pain: Case Series on Knee Osteoarthritis and Updated Review of the Underlying Anatomy and Available Techniques. Biomed Res Int. 2022 May 31;2022:2685898. doi: 10.1155/2022/2685898. eCollection 2022. PMID 35686229
- [Background] Leite CBG, Merkely G, Charles JF, Lattermann C. From Inflammation to Resolution: Specialized Pro-resolving Mediators in Posttraumatic Osteoarthritis. Curr Osteoporos Rep. 2023 Dec;21(6):758-770. doi: 10.1007/s11914-023-00817-3. Epub 2023 Aug 24. PMID 37615856
- [Background] 1. Байбусунова А, Нысанбай Г, Шварц Д, Жакеева М. Diagnosis and treatment of knee osteoarthritis: Modern aspects. J Orthop Trauma. 2024;48(12):21-9.